CLINICAL TRIAL: NCT02968693
Title: Drug Delivery Devices for Osteomyelitis
Status: Completed | Type: Observational
Sponsor: Yulin Orthopedics Hospital of Chinese and Western Medicine (Other)
Responsible Party: Principal Investigator, Shanchao Luo, Director, Yulin Orthopedics Hospital of Chinese and Western Medicine
Other Study IDs: 20150801c
Record Dates: First submitted 2016-11-01; First posted 2016-11-18 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Osteomyelitis
MeSH Terms: conditions — Osteomyelitis | interventions — Vancomycin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- combination therapy group: antibiotic-loaded calcium sulfate and antibiotic-loaded polymethyl methacrylate (PMMA) and Vancomycin
  Interventions: Device: antibiotic-loaded calcium sulfate; Device: antibiotic-loaded polymethyl methacrylate; Drug: Vancomycin
- PMMA group: antibiotic-loaded polymethyl methacrylate and Vancomycin
  Interventions: Device: antibiotic-loaded polymethyl methacrylate; Drug: Vancomycin

INTERVENTIONS:
Device: antibiotic-loaded calcium sulfate — To obtain a paste suitable for pellets, the following steps should be used: 1. Empty 10 cc Stimulan® calcium sulfate powder (Stimulan; Biocomposites Ltd; United Kingdom) into a sterile mixing bowl. 2. The calcium sulfate powder was mixed with 2,000 mg of vancomycin powder. 3. Add approximately 5 ml mixing solution into the above mixture. Mix thoroughly until a smooth paste is formed (approximately 30 seconds). 4. The resultant paste is uniformly smooth into the mould provided to form pellets with diameters of 4.8 mm and height of 3.3 mm. 5. Allow paste to cure undisturbed for at least 15 minutes after mixing. Flex mould to release pellets.
  Groups: combination therapy group
Device: antibiotic-loaded polymethyl methacrylate — One sachet of 40g PALACOSR®+G power containing 33.6g PMMA and with the addition of 0.5g gentamicin sulphate (Heraeus Medical Gesellschaft mit beschränkter Haftung,Germany) was mixed with 4,000 mg of vancomycin powder in a sterile bowl. The liquid provided was poured into the resultant mixture above. Then, the mixture was stirred carefully for 30 sec. If the dough-like mass no longer sticked to the rubber gloves, it can be progressed. If the required consistency was obtained, the cement can be applied to the bony defect until it hardened completely.
Drug: Vancomycin — Vancomycin powder was added into the combination therapy group and PMMA groups

SUMMARY:
Fifty-one patients suffering from chronic post-traumatic or postoperative osteomyelitis of the lower extremities were included in the retrospective investigation. The patients were assigned to the study group of the combination therapy with antibiotic-loaded calcium sulfate and antibiotic-loaded PMMA or the control group of the antibiotic-loaded PMMA. Hematological parameters, eradication of infection, rate of infection recurrence and reoperation rate were evaluated during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The retrospective study included patients with chronic post-traumatic or postoperative osteomyelitis and excluded patients suffering from hematogenous osteomyelitis or acute post-traumatic or postoperative osteomyelitis.

Exclusion Criteria:

* Other kinds of osteomyelitis.

Ages: 15 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between April 2011 and April 2015, fifty-one patients requiring surgical treatment for chronic post-traumatic/postoperative osteomyelitis of the lower extremities were enrolled in a retrospective and control study in our hospital.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2011-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
complications after first-stage surgery. | through study completion, an average of 24 months.
local infection recurrence after first-stage surgery. | through study completion, an average of 24 months.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Yulin Orthopedics Hospital of Chinese and Western Medicine, Yulin, Guangxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo S, Jiang T, Yang Y, Yang X, Zhao J. Combination therapy with vancomycin-loaded calcium sulfate and vancomycin-loaded PMMA in the treatment of chronic osteomyelitis. BMC Musculoskelet Disord. 2016 Dec 22;17(1):502. doi: 10.1186/s12891-016-1352-9. PMID 28007027